CLINICAL TRIAL: NCT06204588
Title: Clinical and Radiographic Evaluation of Volume Stable Collagen Matrix (VCMX) in the Regenerative Outcome of Periodontal Horizontal Bone Loss When Used With Diode Laser Therapy in Humans: A Randomized Controlled Clinical Trial
Brief Title: Evaluation of Regenerative Potential in Horizontal Bone Loss Using VCMX Along With LASER Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shikha IMRG Perio
Record Dates: First submitted 2023-12-14; First posted 2024-01-12 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Bone Loss, Alveolar
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test group-1 (Experimental): using collagen matrix and laser therapy in horizontal bone loss defects by single flap approach (SFA+VCMX+LLLT).
  Interventions: Procedure: Test group 1: VCMX + Low level LASER therapy + Single flap approach
- Test group-2 (Experimental): Single flap approach along with diode laser (SFA+LLLT).
  Interventions: Procedure: Test group 2: Low level LASER therapy + Single flap approach
- Control group (Experimental): using single flap approach only
  Interventions: Procedure: control group: SFA only

INTERVENTIONS:
Procedure: control group: SFA only — Single flap approach
  Arms: Control group
Procedure: Test group 1: VCMX + Low level LASER therapy + Single flap approach — using collagen matrix and laser therapy in horizontal bone loss defects by single flap approach (SFA+VCMX+LLLT).
  Arms: Test group-1
Procedure: Test group 2: Low level LASER therapy + Single flap approach — Laser therapy in horizontal bone loss defects by single flap approach (SFA+LLLT).
  Arms: Test group-2

SUMMARY:
Background- Periodontitis, an inflammatory disease of the periodontium, is one of the major causes of tooth mortality. Of all the bone destruction patterns that are present in periodontitis, horizontal bone loss is the most common. Therefore, treatment modalities that help in rebuilding horizontal defects are vital in total periodontal reconstruction.

Rationale- The supracrestal bone regeneration in cases of horizontal bone loss has remained a mirage with very little recorded success. Volume stable collagen matrix(VCMX), is a porous, cross-linked collagen matrix of porcine origin designed to facilitate cell and vascular ingrowth and soft-tissue volume augmentation, may be beneficial in maintaining the supracrestal space and may overcome the limitation of bone regeneration in horizontal defects. Evidence has shown that Low level laser therapy(LLLT) based on principal of biostimulation of osteoclastic cells, can have a positive effect on the regeneration of supracrestal bone in horizontal bone destruction. So, this study will be first of its kind using combination of VCMX with LLLT to assess regenerative outcome in treatment of horizontal bone destruction in patients with periodontitis.

Objectives: To assess clinical and radiographic regenerative outcome of periodontal tissues using LLLT and placing VCMX with single flap approach(SFA) in treatment of horizontal bone loss as compared to LLLT and SFA.

Method: A total of 60 patients will be randomly divided into three groups: Test Group 1: VCMX +LLLT +SFA, Test Group 2:LLLT+SFA, and Control group: SFA. Periodontal parameters will be evaluated at baseline, 3, 6, and 9 months. CBCT will be evaluated at baseline and 9 months.

Expected outcome: VCMX with Laser could achieve supracrestal bone regeneration in horizontal bone loss.

DETAILED DESCRIPTION:
Periodontitis is a chronic inflammatory disease triggered by gram-negative anaerobic microbes and involves chronic inflammation that causes the destruction of the tooth-supporting apparatus and can lead to tooth loss.1 Periodontal disease is responsible for decreasing alveolar bone height along with morphologic changes of alveolar bone. Various pattern of bone loss was observed clinically horizontal and vertical pattern of bone loss are most commonly seen in periodontitis cases.2 Various factors that determine bone loss patterns are teeth alignments in arch root position within the alveolar socket and root proximity with the adjacent tooth surface.3 Kern et al in 1984 called this horizontal bone defect as zero wall defects. In this type of defect bone margin reduction occurs horizontally and its margin lies perpendicular to tooth surface. Horizontal pattern of bone loss is most commonly seen in human dentition4 but it receives very less attention in terms of treatment modalities. The prevalence of vertical bone loss was 7.8% with treatment choices of 96.8% while the horizontal bone loss prevalence rate was 92.2% and undergo 3.2% treatment options only.5 Due to no bone wall remaining for the support and stability of grafts and membranes, leads to a very low success rate of horizontal bone defects treatment modalities. To regenerate the lost part of the alveolar bone is always a challenge for both clinician and patient.

Several attempts have been done for the treatment of horizontal bone defects using bone grafts, membranes, or a combination of grafts and membranes. Recently recombinant human bone morphogenic protein (rhBMP) and enamel matrix proteins(EMPs) have been assessed for the management of horizontal defects. But their results were mixed and sometimes disappointing. The single flap approach (SFA) is a simplified minimally invasive surgical approach that enhances primary closure and minimizes tissue trauma. The principle behind using this approach is that elevation of the limited mucoperiosteal flap allows surgical access from either the buccal or palatal/lingual aspect only depending on the extension of the lesion, leaving the interdental supracrestal gingival tissue intact. Main advantages associated with this approach that flap repositioning and suturing to the undetached papilla, thereby preventing contamination by blood clots and reduction in post-surgical reduction. Due to the emergence of biologic approach and biomaterials there is improved concern toward of horizontal defects. Various factors determine the outcomes like patient-related factors, site-related and clinician related factors. Laser technology now a days becoming popular in various medical applications like photodynamic therapy. Low level laser therapy (LLLT) also called photo-biomodulation enhance wound healing based on the principle of biomodulatory capacity of laser on body cells leading to increased cell activity.12 It reduces excessive post-operative inflammation, edema and pain. LLLT can promote bone regeneration by enhancing proliferation and differentiation of human osteoblasts.14 According to Gavish et al 780nm diode laser shown to inhibit the gene expression of pro-inflammatory cytokines interleukin-1 beta(IL-1β) ,modulate matrix metalloproteinase (MMPs) activity15 and reduce monocyte chemotactiprotein-1 (MCP-1), IL-1α, IL-10 and IL-6 in lipopolysaccharide-stimulated macrophages.16 Numerous treatment approaches for restoring such defects have been investigated. Despite laudable record, autografts have been questioned for surgical invasiveness, donor site morbidity, limited quantity of donor material and increased operating time for harvesting procedures.17 Limitations of the use of osteoinductive grafts is variation in bone induction capacity sourced from different tissue banks.18,19 When used in intrabony defects, Enamel Matrix Derivative(EMD) may restrict the space provision potential of the preparation.20 Further, application of EMD is a technique sensitive procedures and contamination of the material jeopardizing the regenerative potential. The lack of rigidity and rapid degradation (biodegradability) make the use of PRF for periodontal regeneration difficult. Nanocomposites and nanostructured materials are thought to have a key function in hard tissue research, since natural bone tissue is a distinctive model of a nanocomposite. Collagen has been potentially used in periodontal tissue engineering. The integration of collagen as a structural protein, serving as an essential component of connective tissue into three-dimensional scaffolds implanted after periodontal injury, necrosis or inflammation has attracted much attention in tissue regeneration.

According to Ibara et al, scaffolds to be implanted are durable if composed of nanoparticles. The nanoparticles facilitate healing process in contact with the tissues intended for the reformation. Recently, Thoma et al developed and tested collagen-based matrices as potential devices for soft tissue volume augmentation. Volume stable collagen matrix (VCMX) is able to overcome the volume stability limitation of most commercially available grafts.21 It is one of the most biocompatible, novel material to be used in this study. While mechanical stability is achieved by chemical crosslinking, mechanical testing demonstrated preserved elasticity of the material over 14 days.22 It has shown quite impressive results in resolving the intrabony defects in animal studies with an average of 58.56% of new bone formation .23 Imber J-C et al23, preclinically evaluated the effect of a volume-stable collagen matrix on periodontal regeneration in two-wall intrabony defects. This study provided histologic evidence for the potential of this novel VCMX to facilitate periodontal regeneration. Asparuhova, M.B et al24 investigated the influence of a novel volume-stable collagen matrix (VCMX) on early wound healing events including cellular migration and adhesion, protein adsorption and release, and the dynamics of the hemostatic system. Their study concluded that their data strongly support the effect of the novel VCMX on fibrin clot stabilization and coagulation/fibrinolysis equilibrium, thus facilitating progression to the next stages of the soft tissue healing process.

Therefore, the present study was planned to evaluate the supracrestal regenerative potential of volume stable collagen matrix (VCMX) along with single flap approach(SFA) when used with diode laser in the treatment of horizontal bone defect of stage 2 and 3 patients in comparison to OFD with diode laser and OFD alone.

Methodology:

* Study design and settings: The study design is "Randomized controlled clinical trial" and will be conducting in Department of Periodontology, Post graduate Institute of Dental Sciences, Rohtak, Haryana.
* Study population:

Systemically healthy patients with periodontitis stage 2 and stage 3 having horizontal bone loss will be enrolled in the present study.

I Study conduct: Patients will be enrolled according to inclusion and exclusion criteria from the outpatient department of periodontics, Post Graduate Institute of Dental Sciences, Rohtak, Haryana. Informed and written consent will be taken from each patient in his or her language.

Randomization of patients would be done by generating the allocation sequence using computer-generated table by another investigator. Patients will be randomly allocated into:

* Control group: using single flap approach only
* Test group 1: using collagen matrix and laser therapy in horizontal bone loss defects by single flap approach (SFA+VCMX+LLLT).
* Test group 2: Single flap approach along with diode laser (SFA+LLLT). A balanced, permuted block approach (in blocks of four and six patients) will be used to prepare the randomization tables. After the debridement of the bone defect, the eligibility of the bone defect would be confirmed. Allocation concealment will be performed by opaque sealed envelopes that would be opened after debridement of horizontal bone loss defects, and the surgeon will be informed of the allocated treatment. Although the surgeon won't be blinded to the treatments, the examiners recording clinical and radiographic parameters would be blind to the treatment groups. Minimum One horizontal bone defect per patient will be included in the study.

Periodontal parameters:

Parameters recorded for experimental and adjacent teeth will include: PIaque index (PI) and Gingival Index (GI), assessed at six surfaces (mesiobuccal, midbuccal, distobuccal, midlingual/midpalatal, mesiolingual, distolingual); bleeding on probing (BOP, %), PPD, CAL, and gingival recession (REC), examined at six surfaces (mesiobuccal, midbuccal, disto-buccal, mesiolingual/mesiopalatal, midlingual/midpalatal, distolingual/distopalatal).

Radiographic Parameters that will be assessed using CBCT will include alveolar crest changes (ACC).Outcome measures will be revaluated at 3, 6, & 9 months interval

Intervention:

Presurgical patient preparation:

Patients diagnosed with periodontitis who will meet the inclusion criteria will be screened for periodontal examination. Based on this examination, target sites will be identified. Each patient will receive the initial phase of the therapy, which will include oral hygiene instructions, supragingival and subgingival debridement using ultrasonic (Piezon®, EMS Dental, Nyon, Switzerland) and hand instrumentations (Gracey Curettes,Hu- Friedy®, Chicago, IL, USA), and relieving of occlusal trauma.

Surgical procedure:

Surgical sites will be anaesthetized using local anaesthesia. Simplified Papilla Preservation flap technique will be exercised using single flap approach. Crevicular incisions will be made on buccal/lingual/palatal sites to raise a full-thickness mucoperiosteal flap. Precaution would be taken to preserve the maximum interdental gingival tissue at the time of crevicular incision, and no bone recontouring would be performed. Thorough debridement of the surgical site would be performed For the test group1, VCMX would be placed according to the dimensions of the horizontal bone loss defect along with the use of diode laser (LLLT) on the inner epithelium of flap. For the test group 2, SFA will be done along with the use of diode laser (LLLT). For control group, SFA will be done. And after this, flap would be approximated and sutured at the original position with a monofilament suture material using interrupted sutures.

Instructions for maintenance of proper oral hygiene will be reinforced. Study participants will be scheduled for a follow-up visit weekly to1-month postsurgery and subsequently at 3-, 6-, and 9-month intervals.

All statistical tests will use two-sided P values, and statistical software will be used in the analysis of the study data. Differences associated with P values 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Periodontitis stage 2 and stage 3 patients will be enrolled according to criteria of 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions
* Horizontal bone loss defects with depth ≥ 5 mm (initially analyzed by trans-gingival probing and intraoral periapical radiographs and will be confirmed further after flap elevation and CBCT)
* PPD ≥ 5 mm
* CAL ≥ 3 mm
* Tooth mobility < grade 1
* Experimental teeth and adjacent teeth would be required to be vital and free of caries or dental restorations

Exclusion Criteria:

* Any systemic illness that could affect the periodontium or outcome of periodontal therapy
* patients on medications such as corticosteroids or calcium channel blockers
* long-term nonsteroidal anti-inflammatory drug therapy
* pregnant or lactating women
* current and past smoker
* Periodontitis stage 4
* teeth with one-wall defect, the presence of exostoses and ledges, grade II and grade III mobile teeth, defects extending to a root furcation area, unrestorable teeth, fractured/perforated roots, developing permanent teeth, endodontically treated teeth, and teeth with premature contact and dental prosthesis.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level | 24 months
  Periodontal probe will be used to measure clinical attachment level
alveolar bone level | 24 months
  transgingival probing using periodontal probe and by radiographically using CBCT

CONTACTS AND LOCATIONS:
Overall Officials: Shikha Tewari, Principal Investigator — Post graduate institute of Dental Sciences ROHTAK
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No